CLINICAL TRIAL: NCT06561997
Title: Enhancing Thoracolumbar Burst Fracture Treatment: The Advantage of Robot-Assisted Posterior Fixation for Improved Reduction and Collapse Prevention
Brief Title: Enhancing Thoracolumbar Burst Fracture Treatment
Status: Completed | Type: Observational
Sponsor: Peng Liu (Other)
Responsible Party: Sponsor-Investigator, Peng Liu, Professor, Sichuan Provincial People's Hospital
Organization: Sichuan Provincial People's Hospital (Other)
Other Study IDs: 2024-42
Record Dates: First submitted 2024-07-19; First posted 2024-08-20 (Actual); Last update posted 2024-08-20 (Actual); Status verified 2024-08

CONDITIONS: Surgery
Keywords: Thoracolumbar fractures; Percutaneous pedicle screw fixation; Robot-assisted; Endplate collapse
MeSH Terms: interventions — Robotic Surgical Procedures

STUDY DESIGN:
Observational Model: Case-Control | Time Perspective: Retrospective
Oversight: Data Monitoring Committee: No | FDA-regulated Drug: No | FDA-regulated Device: No

GROUPS / COHORTS (2):
- Robot-assisted group: received percutaneous pedicle screw fixation (PPSF) with robotic assistance
  Interventions: Device: Robot-assisted
- Free-hand group: received percutaneous pedicle screw fixation (PPSF) without robotic assistance
  Interventions: Device: Free-hand

INTERVENTIONS:
Device: Robot-assisted — received percutaneous pedicle screw fixation (PPSF) with robotic assistance
  Groups: Robot-assisted group
Device: Free-hand — received percutaneous pedicle screw fixation (PPSF) without robotic assistance
  Groups: Free-hand group

SUMMARY:
The optimal treatment for neurologically intact thoracolumbar fractures remains controversial. Percutaneous pedicle screw fixation (PPSF) has been proposed for these fractures; however, achieving satisfactory reduction can be challenging. This study applied robot-assisted PPSF to enhance treatment outcomes.

DETAILED DESCRIPTION:
The optimal treatment for neurologically intact thoracolumbar fractures remains controversial. Percutaneous pedicle screw fixation (PPSF) has been proposed for these fractures; however, achieving satisfactory reduction can be challenging. This study applied robot-assisted PPSF to enhance treatment outcomes. The investigators retrospectively analyzed the medical records of 182 consecutive patients with thoracolumbar burst fractures treated with PPSF, with (n=88) and without (n=94) robotic assistance, at our hospital between April 2017 and June 2019. The participants were evaluated surgical time, intraoperative bleeding, radiation dosage, accuracy of screw placement, fractured vertebral height, Cobb's angle, surgery efficacy (pain relief and limb function), and implant failure to assess the potential advantages of robot-assisted PPSF. Robot-assisted PPSF for thoracolumbar burst fractures reduces surgery time and intraoperative bleeding, enhances screw placement accuracy, and achieves better reduction compared to the free-hand technique. This approach effectively prevents endplate collapse and recurrence of kyphosis post-surgery. However, functional recovery in the short term is similar between the two methods.

ELIGIBILITY:
Inclusion Criteria:

had thoracolumbar burst fractures classified as Magerl type A3 underwent short segment posterior fixation (SSPF) showed no signs of osteoporosis on dual-energy X-ray absorptiometry in patients older than 60 years.

Exclusion Criteria:

had fractures outside the T11-L2 range presented with old fractures, (iii) had a Parker score ≥ 7 had multiple segment fractures had neurological deficiency caused by fractures had concomitant pain caused by spinal degeneration such as lumbar disc protrusion, spondylolisthesis, spinal stenosis, and/or scoliosis could not receive pedicle screw placement due to bilateral pedicle fractures with displacement had incomplete clinical data or were lost to follow-up

Ages: 18 Years to 64 Years | Sex: All | Healthy Volunteers: No
Age Groups: Adult
Study Population: The investigators retrospectively analyzed the medical records of 182 consecutive patients (142 men, 40 women; average age: 38.8 years, age range: 18-64 years) with thoracolumbar burst fractures who had received percutaneous pedicle screw fixation (PPSF) with or without robotic assistance at our hospital between April 2017 and June 2019. The causes of trauma were falls from height (94 patients), traffic accidents (70 patients), and heavy object strikes (18 patients). The time elapsed from fracture occurrence to surgery ranged from 1 to 7 days (average: 2.4 days). The fractures were located at the T11 level in 36 patients, T12 in 73, L1 in 58, and L2 in 15.
Sampling Method: Non-Probability Sample
Enrollment: 182 (Actual)
Dates: Start 2017-04-01 (Actual); Primary Completion 2019-06-30 (Actual); Study Completion 2020-06-30 (Actual)

PRIMARY OUTCOMES:
The height of sagittal kyphosis | One week post-surgery
  The height of sagittal kyphosis of the injured vertebral body
The Cobb's angle of sagittal kyphosis | One week post-surgery
  The Cobb's angle of sagittal kyphosis of the injured vertebral body
The height of sagittal kyphosis | One-year post-surgery
  The height of sagittal kyphosis of the injured vertebral body
The Cobb's angle of sagittal kyphosis | One-year post-surgery
  The Cobb's angle of sagittal kyphosis of the injured vertebral body

SECONDARY OUTCOMES:
Visual Analogue Scale (VAS) score | One week post-surgery
  Visual Analogue Scale (VAS; out of a total score of 10, 0 corresponds to no pain and 10 refers to unbearable pain)
Visual Analogue Scale (VAS) score | One-year post-surgery
  Visual Analogue Scale (VAS; out of a total score of 10, 0 corresponds to no pain and 10 refers to unbearable pain)
Oswestry Disability Index (ODI) score | One week post-surgery
  Oswestry Disability Index (ODI; the questionnaire is composed of 10 aspects for pain, self-care, extraction, walking, sitting, standing, sleeping, sexual life, social life, and tourism, with 0-5 points for each item. 0% scores corresponded to normal function and 100% corresponded to severe dysfunction)
Oswestry Disability Index (ODI) score | One-year post-surgery
  Oswestry Disability Index (ODI; the questionnaire is composed of 10 aspects for pain, self-care, extraction, walking, sitting, standing, sleeping, sexual life, social life, and tourism, with 0-5 points for each item. 0% scores corresponded to normal function and 100% corresponded to severe dysfunction)

CONTACTS AND LOCATIONS:
Overall Officials: Fei Wang, M.D., Principal Investigator — Sichuan Provincial People's Hospital
Locations (1):
- "Tianji" 3rd generation orthopedic robot, Chengdu, Sichuan, China

IPD SHARING:
Plan to Share IPD: No

REFERENCES:
- [Result] Defino HL, Canto FR. Low thoracic and lumbar burst fractures: radiographic and functional outcomes. Eur Spine J. 2007 Nov;16(11):1934-43. doi: 10.1007/s00586-007-0406-y. Epub 2007 Jun 14. PMID 17566793
- [Result] Kapoen C, Liu Y, Bloemers FW, Deunk J. Pedicle screw fixation of thoracolumbar fractures: conventional short segment versus short segment with intermediate screws at the fracture level-a systematic review and meta-analysis. Eur Spine J. 2020 Oct;29(10):2491-2504. doi: 10.1007/s00586-020-06479-4. Epub 2020 Jun 11. PMID 32529525
- [Result] Aono H, Ishii K, Tobimatsu H, Nagamoto Y, Takenaka S, Furuya M, Chiaki H, Iwasaki M. Temporary short-segment pedicle screw fixation for thoracolumbar burst fractures: comparative study with or without vertebroplasty. Spine J. 2017 Aug;17(8):1113-1119. doi: 10.1016/j.spinee.2017.03.022. Epub 2017 Mar 31. PMID 28373079
- [Result] Scholl BM, Theiss SM, Kirkpatrick JS. Short segment fixation of thoracolumbar burst fractures. Orthopedics. 2006 Aug;29(8):703-8. doi: 10.3928/01477447-20060801-14. PMID 16924864
- [Result] Magerl F, Aebi M, Gertzbein SD, Harms J, Nazarian S. A comprehensive classification of thoracic and lumbar injuries. Eur Spine J. 1994;3(4):184-201. doi: 10.1007/BF02221591. PMID 7866834